CLINICAL TRIAL: NCT02475746
Title: A Phase 1, Open-label, Two-period, Fixed-sequence Study To Estimate The Effects Of Multiple-dose Administration Of Itraconazole On The Single-dose Pharmacokinetics Of Pf-06372865 In Healthy Adult Subjects
Brief Title: An Open-label, Two-period, Fixed-sequence Study to Evaluate Multiple-dose Itraconazole Effect on The Single-dose PK of PF-06372865 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7431009
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: drug interaction, PF-06372865, itraconazole
MeSH Terms: interventions — PF-06372865; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06372865 treatment arm (Experimental): treatment arm includes two treatment periods, a single dose of PF-06372865 (period 1) followed by 8-days itraconazole with a single dose of PF-06372865 co-administered on Day 4
  Interventions: Drug: PF-06372865; Drug: itraconazole

INTERVENTIONS:
Drug: PF-06372865 — single dose of 7.5 mg PF-06372865 alone (period 1) or co-administered with itraconazole (period 2)
Drug: itraconazole — Interacting drug which will be given 200 mg QD for 8 days in period 2

SUMMARY:
The purpose of this study is to evaluate the effect of itraconazole after multiple dose administration on the single dose PK of PF-06372865.

DETAILED DESCRIPTION:
Study includes two treatment periods: period 1 is single dose of PF-06372865 given alone followed by at least 5-day washout out. The period 2 is 200 mg QD itraconazole given for 8 days with PF-06372865 single dose co-administered on day 4 (1 hour later than itraconazole dose). The PK and safety will be assessed and compared for single dose of PF-06372865 in period 1 and period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects who, at the time of Screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Hypersensitivity or previous adverse events due to azole antifungals.
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Use of tobacco or nicotine containing products in the past 6 months, as evident by a positive urine Cotinine test at Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement or 5 half-lives preceding the first dose of investigational product, whichever is longer.
* Screening supine blood pressure 140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Screening supine 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at Screening.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at Screening AND at Day 0, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary: Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) >1x upper limit of normal (ULN); Total bilirubin >1x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ULN.
* Pregnant female subjects; females of childbearing potential; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least two months after the last dose of Itraconazole
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor. Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of investigational product
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study
* Any condition possibly affecting drug absorption (eg, gastrectomy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Cmax ratio of PF-06372865 alone vs coadministration with itraconazole | 0 to 120 hours post PF-06372865
  The ratio of maximum plasma concentration of PF-06372865 following single dose co-administered with itraconazole vs given alone
AUC ratio of PF-06372865 alone vs coadministration with itraconazole | 0 to 120 hours post PF-06372865
  The ratio of AUC (area under plasma concentration curve) of PF-06372865 following single dose co-administered with itraconazole vs given alone
PF-06372865 Tmax | 0 to 120 hours post PF-06372865
  Time to PF-06372865 maximum concentration following single dose co-administered with itraconazole or given alone
T1/2 of PF-06372865 alone vs coadministration with itraconazole | 0 to 120 hours post PF-06372865
  T1/2 (half-life) of PF-06372865 following single dose co-administered with itraconazole or given alone
CL/F of PF-06372865 alone vs coadministration with itraconazole | 0 to 120 hours post PF-06372865
  CL/F (oral clearance) of PF-06372865 following single dose co-administered with itraconazole or given alone
Vz/F of PF-06372865 alone vs coadministration with itraconazole | 0 to 120 hours post PF-06372865
  Vz/F (volume distribution) of PF-06372865 following single dose co-administered with itraconazole or given alone

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer New Haven Clinical Research Unit, New Haven, Connecticut
  - CRU New Haven, New Haven, Connecticut